CLINICAL TRIAL: NCT00727532
Title: Correlation of Pathologic Findings After Neo-adjuvant Sorafenib With Results of Diffusion-Weighted Magnetic Resonance Imaging in Patients With Locally Advanced or Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Sorafenib in Treating Patients With Locally Advanced or Metastatic Kidney Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 07U1; P30CA060553 (NIH); NU-IRB-STU00003123 (Other: Northwestern University IRB)
Record Dates: First submitted 2008-08-01; First posted 2008-08-04 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2018-10

CONDITIONS: Hereditary Clear Cell Renal Cell Carcinoma; Kidney Cancer
Keywords: clear cell renal cell carcinoma; hereditary clear cell renal cell carcinoma; recurrent renal cell cancer; stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): Eligible patients undergo pre-treatment DW-MRI of the abdomen and pelvis. Patient then receive Sorafenib 400mg orally twice daily on days 1-28. Following completion of 28 days of sorafenib, patients obtain a second DW-MRI.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 400mg by mouth twice daily for 28 consecutive days
  Other Names: Nexavar

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sorafenib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying how well sorafenib works in treating patients with locally advanced or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To demonstrate the feasibility and safety of sorafenib tosylate when given prior to nephrectomy or metastasectomy.
* To evaluate the ability of diffusion-weighted magnetic resonance imaging (DW-MRI) to detect early and ongoing microstructural changes in primary and metastatic renal cell carcinoma lesions during neoadjuvant therapy with sorafenib tosylate.
* To correlate early and ongoing microstructural changes in primary and metastatic renal cell carcinoma lesions with pathologic and clinical findings at the time of nephrectomy or metastasectomy.
* To evaluate the ability of changes in DW-MRI to predict subsequent favorable response to treatment (complete or partial response or stable disease) after 4 weeks of therapy.

OUTLINE: Patients receive oral sorafenib tosylate twice daily on days 1-28. Patients then undergo a nephrectomy or metastasectomy in week 5. Patients with residual metastatic disease may continue sorafenib tosylate twice daily and undergo a diffusion-weighted MRI (DW-MRI) every 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo a DW-MRI of the abdomen and pelvis at baseline and prior to week 5 to evaluate microstructure tumor changes and to allow for prediction of sorafenib tosylate benefit. DW-MRI results are correlated with surgical and pathologic findings obtained at week 5.

Resected tumor tissue are analyzed for vascular density and to distinguish apoptotic cell death from necrotic cell death via immunohistochemistry and to measure apoptotic cell death via TUNEL assay.

After completion of study treatment, patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed clear cell renal cell carcinoma, meeting 1 of the following criteria:

  * Localized disease, as evidenced by intact, bulky, and primary renal lesions (T1 > 3 cm, any T2, T3, or T4) appropriate for nephrectomy
  * Limited metastatic disease, as evidenced by any renal primary (T1 > 3 cm, any T2, T3, or T4) appropriate for cytoreductive nephrectomy
  * Isolated abdominal/pelvic recurrence with limited metastatic burden (minimum size > 2 cm) appropriate for metastasectomy
* No known brain metastasis

  * Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group performance status 0-1
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alanine aminotransferase and Aspartate aminotransferase ≤ 2.5 times ULN (≤ 5 times ULN with liver involvement)
* Creatinine ≤ 1.5 times ULN
* Estimated glomerular filtration rate > 30 mL/min (for patients receiving Gd-enhanced MRI)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during (men and women), and for at least 3 months after (men) completion of study therapy
* Adequate cardiac and pulmonary status for operative therapy
* No active clinically serious infection > CTCAE grade 2
* No known HIV, hepatitis B, or hepatitis C infections
* No serious non-healing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 4 weeks
* No pulmonary hemorrhage/bleeding event ≥ CTCAE grade 2 within the past 4 weeks
* No other hemorrhage/bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* No history of an uncontrolled bleeding disorder including, but not limited to, any of the following:

  * Bleeding diathesis
  * Coagulopathy
* No cardiac disease or condition including, but not limited to, any of the following:

  * New York Heart Association class II-IV congestive heart failure
  * Unstable angina (anginal symptoms at rest)
  * New onset angina beginning within the last 3 months
  * Myocardial infarction within the past 6 months
  * Cardiac ventricular arrhythmias requiring antiarrhythmic therapy
* No uncontrolled hypertension (i.e., systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 100 mm Hg) despite optimal medical management
* No thrombolic or embolic events within the past 6 months (e.g., cerebrovascular accident including transient ischemic attacks)
* No condition that impairs the ability to swallow whole pills
* No malabsorption problem
* No contraindication to MRI, including, but not limited to, any of the following:

  * Ferromagnetic implants
  * Dental work
  * Pacemakers
  * Metallic implants
  * Severe claustrophobia which precludes closed MRI testing
* No known or suspected allergy to sorafenib tosylate
* No contraindication or allergy to gadolinium (e.g., end stage renal disease requiring hemodialysis)
* No intercurrent illness or situation which, in the judgment of the investigator, would affect assessments of clinical status and study endpoints significantly

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior major surgery or open biopsy
* No prior therapy with tyrosine kinase or vascular endothelial growth factor inhibitors (e.g., sunitinib malate, sorafenib, or bevacizumab)
* No concurrent Hypericum perforatum (St. John's wort) or rifampin
* No concurrent use of illicit drugs or other substances that may, in the opinion of the investigator, have a reasonable chance of contributing to toxicity or interfering with study results

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open to enrollment at Northwestern University beginning June 2008, and closed to enrollment in September 2012.
Groups:
- Sorafenib: Sorafenib 400mg orally twice daily on days 1-28
  sorafenib tosylate: 400mg by mouth twice daily for 28 consecutive days
  diffusion-weighted magnetic resonance imaging: At baseline and just prior to surgery after sorafenib treatment
Period: Overall Study
Arm/Group | Sorafenib
Started | 9
Completed | 7
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Sorafenib: Sorafenib 400mg orally twice daily on days 1-28
Arm/Group | Sorafenib
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9
Renal cell carcinoma Clinical Staging [Number; unit: participants] — Participants must have bulky (T1>3cm,any T2, T3,orT4) renal cell carcinoma undergoing nephrectomy.Staging defined as:T1>3cm: Tumor ≤7cm in greatest dimension but >3cm, limited to the kidney;T2:Tumor >7cm, limited to the kidney;T3:Tumor extends into major veins but not into the ipsilateral adrenal gland & not beyond Gerota fascia (the fibrous layer that surrounds the kidney & nearby fatty tissue);T4:Tumor invades beyond Gerota fascia(including contiguous extension into ipsilateral adrenal gland).The higher the number after the T, the larger the tumor or more it has grown into nearby tissues.
  participants
    T1>3cm | 0
    T2 | 0
    T3 | 8
    T4 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Difference in Apparent Diffusion Coefficient Between Baseline and Week 5
Description: Mean Difference in Apparent Diffusion Coefficient [Time Frame: Baseline and Week 5] To assess whether changes in the apparent diffusion coefficient (ADC) during neoadjuvant sorafenib treatment are detectable in locally advanced or metastatic kidney cancer. The ADC value will be calculated at baseline (within 28 days of initiating sorafenib) and Week 5, and the mean difference will be calculated. The percent change between this mean difference is reported. Week 5 ADC value minus baseline ADC value/divided by baseline ADC value was calculated for each participant. Apparent diffusion coefficient (ADC), obtained by measuring diffusion values at magnetic resonance imaging (MRI), is a measure of water mobility. Lower values correspond to tumor and higher values are consistent with cysts. With sorafenib therapy, the amount of free water may increase in a lesion due to necrosis, and as a result the ADC may increase in value.
Time Frame: Baseline and week 5
Measure: Mean (Full Range); unit: Percent change
Arm/Group | Sorafenib
Number analyzed (Participants) | 7
Percent change | -7.57 [-59.00 to 49.40]

2. Primary Outcome: Change in Tumor Size From Baseline to Approximately 29-34 Days After Completion of Neoadjuvant Sorafenib Treatment
Description: Tumors were measured at baseline and approximately 29-34 days after completion of neoadjuvant treatment with sorafenib (just prior to surgery). Tumors were assessed by RECIST response criteria.
Time Frame: Just prior to study week 5
Measure: Median (Full Range); unit: percent change
Arm/Group | Sorafenib
Number analyzed (Participants) | 7
percent change | -5.34 [-15.3 to 7.2]

3. Post Hoc Outcome: Percentage Change of Necrosis From Baseline to Surgery
Description: Changes in MRI will be correlated with findings of necrosis. Amount of necrosis will be measured at baseline and at time of surgery. Percentage change for necrosis will be calculated from baseline and time of surgery.
Time Frame: At time of surgery
Measure: Mean (Full Range); unit: Percentage change
Arm/Group | Sorafenib
Number analyzed (Participants) | 7
Percentage change | 20.13 [-38.32 to 92.92]

ADVERSE EVENTS:
Time Frame: Adverse events assessed for 28 days prior to surgical resection
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (N=9)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=9)
Mucositis/Stomatitis (functional symptomatic) - Oral Cavity (Gastrointestinal disorders) | 2
Elevated Transaminitis (Investigations) | 2 — alanine aminotransferase, aspartate aminotransferase, or both
Rash (Skin and subcutaneous tissue disorders) | 5
Hand-Foot Skin reaction (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Pain (General disorders) | 1
Fatigue (General disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Elevated creatinine (Investigations) | 2
Fever (General disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Lymphopenia (Investigations) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
The trial did not reach the original goal of 10 subjects. Only 9 out of 10 patients had been enrolled, with no accrual for a period of more than 1 year. Therefore it was administratively closed by the Data Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes